CLINICAL TRIAL: NCT00539032
Title: Evaluation of the Response to a Single Dose of Menactra® in Children Aged 5 to 8 Years Who Had Previously Received Two Doses of Quadrivalent (A, C, Y, W-135) Meningococcal Polysaccharide Vaccine Before Age 2 Years in Saudi Arabia
Brief Title: Immunology and Safety of Menactra® in Children in Saudi Arabia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA47
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Results first posted 2011-01-24 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Meningitis; Meningococcemia
Keywords: N. meningitidis; Meningitis; Meningococcemia
MeSH Terms: conditions — Meningitis; Meningococcal Infections

ARMS (2):
- Group 1: Menactra® Booster Group (Experimental): Participants who had received 2 doses of quadrivalent (A, C, Y, and W-135) meningococcal polysaccharide vaccine before age 2 years received a booster vaccination with Menactra® vaccine.
  Interventions: Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate
- Group 2: Menactra® Primary Vaccine (Control) Group (Experimental): Participants who had not previously been given any meningococcal vaccine (meningococcal vaccine naive) received a primary vaccination with Menactra® vaccine.
  Interventions: Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate

INTERVENTIONS:
Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra® Vaccine
  Arms: Group 1: Menactra® Booster Group
Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra® Vaccine
  Arms: Group 2: Menactra® Primary Vaccine (Control) Group

SUMMARY:
This study will be conducted among children in Saudi Arabia who previously received two doses of A, C, Y, W-135 polysaccharide vaccine before the age of 2 years, and in meningococcal vaccine-naïve children (Control Group). This study will evaluate the administration of Menactra® in terms of the serum bactericidal antibody it induces in the two study groups. Safety of Menactra® vaccine will be described.

ELIGIBILITY:
Inclusion Criteria :

* Healthy, as determined by medical history and physical examination.
* Aged between 5 to 8 years on the day of inclusion (from 5th birthday to 1 day before 9th birthday inclusive).
* For the Booster Group , two doses of a quadrivalent (A, C, Y, W-135) meningococcal polysaccharide vaccine received before age 2 years
* For the Control Group , no previous history of any meningococcal vaccination
* Informed consent form signed by the parent(s) or other legal representative
* Able to provide a vaccination log or has available vaccination record in the Health Center.
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria :

* Serious chronic disease (i.e., cardiac, renal, neurologic, metabolic, rheumatologic, psychiatric, etc.)
* Known or suspected impairment of immunologic function.
* Acute medical illness with or without fever within the last 72 hours or a oral temperature ≥ 37.5°C at the time of inclusion.
* Administration of immune globulin or other blood products within the last three months, injected or oral corticosteroids or other immunomodulatory therapy within six weeks of the trial vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial provided that they have not received more than one course within the last two weeks prior to enrollment.
* Oral or injected antibiotic therapy within the 72 hours prior to vaccination.
* Received any vaccine in the 14-day period prior to trial vaccination, or scheduled to receive any vaccination during the 14-day period after trial vaccination.
* Previous history of documented invasive meningococcal disease.
* For the Control Group, previous history of any meningococcal vaccination.
* Systemic hypersensitivity to any of the vaccines components or history of a life-threatening reaction to the trial vaccines or a vaccine containing the same substances.
* Participation in another clinical trial in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Any condition, which, in the opinion of the investigator, would pose a health risk to the subject, or interfere with the evaluation of the vaccine.
* Personal or family history of Guillain Barré syndrome.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (4):
- Saudi Arabia (4):
  - AlKhaleej, Al-Qassim Region
  - AlRabwa, Al-Qassim Region
  - S. Buraida, Al-Qassim Region
  - Safra-Al Midhnab, Al-Qassim Region

REFERENCES:
- [Derived] Khalil M, Al-Mazrou Y, Findlow H, Chadha H, Bosch Castells V, Johnson DR, Borrow R. Safety and immunogenicity of a meningococcal quadrivalent conjugate vaccine in five- to eight-year-old Saudi Arabian children previously vaccinated with two doses of a meningococcal quadrivalent polysaccharide vaccine. Clin Vaccine Immunol. 2012 Oct;19(10):1561-6. doi: 10.1128/CVI.00260-12. Epub 2012 Aug 1. PMID 22855388
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 30 September to 03 November 2007, at 4 health centers in Saudi Arabia.
Pre-assignment Details: A total of 238 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Period: Overall Study
Arm/Group | Group 1: Menactra® Booster Group | Group 2: Menactra® Primary Vaccine (Control) Group
Started | 153 | 85
Completed | 151 | 84
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Menactra® Booster Group | Group 2: Menactra® Primary Vaccine (Control) Group | Total
Number analyzed (Participants) | 153 | 85 | 238
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 153 | 85 | 238
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.12 (0.60) | 6.52 (1.22) | 6.26 (0.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 47 | 131
  Male | 69 | 38 | 107
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 153 | 85 | 238

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Number of Participants Reporting At Least 1 Solicited Injection Site or Systemic Reaction Post-Vaccination With Menactra®
Description: Solicited injection Site reactions: Pain, erythema, and swelling; Solicited systemic reactions: Fever, headache, malaise and myalgia.
Time Frame: Days 0-7 Post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat safety population.
Measure: Number; unit: Participants
Arm/Group | Group 1: Menactra® Booster Group | Group 2: Menactra® Primary Vaccine (Control) Group
Number analyzed (Participants) | 151 | 85
Participants
  Any Solicited Injection Site Reaction | 35 | 19
  Any Pain | 32 | 15
  Grade 3 Pain (Incapacitating) | 1 | 0
  Any Erythema | 10 | 8
  Grade 3 Erythema (≥ 5 cm) | 0 | 0
  Any Swelling | 11 | 8
  Grade 3 Swelling (≥ 5 cm) | 0 | 0
  Any Solicited Systemic Reaction | 36 | 16
  Any Fever | 16 | 8
  Grade 3 Fever (> 39.0 ºC) | 1 | 2
  Any Headache | 13 | 5
  Grade 3 Headache (Prevents daily activities) | 0 | 0
  Any Malaise | 18 | 11
  Grade 3 Malaise (Prevents daily activities) | 0 | 0
  Any Myalgia | 21 | 10
  Grade 3 Myalgia (Prevents daily activities) | 0 | 0

2. Primary Outcome: Geometric Mean Titers (GMTs) as Measured by Serum Bactericidal Assay Using Baby Rabbit Complement (SBA-BR) Pre- and Post-Menactra® Vaccination.
Time Frame: Day 0 (baseline or pre-vaccination) and Day 28 Post-vaccination
Population: Geometric mean titers by serum bactericidal assay were determined in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Menactra® Booster Group | Group 2: Menactra® Primary Vaccine (Control) Group
Number analyzed (Participants) | 140 | 81
Titers
  Serogroup A: Pre-vaccination | 168.9 [117.4 to 243.1] | 196.4 [119.0 to 324.0]
  Serogroup A: Day 28 Post-vaccination | 6991.7 [6107.6 to 8003.8] | 8263.3 [6913.1 to 9877.2]
  Serogroup C: Pre-vaccination | 2.5 [2.2 to 3.0] | 4.1 [2.8 to 5.9]
  Serogroup C: Day 28 Post-vaccination | 167.2 [115.3 to 242.7] | 512.0 [334.4 to 761.2]
  Serogroup Y: Pre-vaccination | 10.2 [6.8 to 15.2] | 12.4 [7.1 to 21.6]
  Serogroup Y: Day 28 Post-vaccination | 2120.2 [1799.0 to 2498.9] | 2558.3 [2015.5 to 3247.3]
  Serogroup W-135: Pre-vaccination | 3.0 [2.4 to 3.8] | 2.7 [2.1 to 3.5]
  Serogroup W-135: Day 28 Post-vaccination | 2387.7 [1950.1 to 2923.5] | 2763.2 [2153.9 to 3544.8]

3. Primary Outcome: Percentage of Participants With ≥ 4-Fold Rise in Titers for the Menactra® Vaccine Serogroups A, C, Y, and W-135.
Time Frame: Day 28 Post-vaccination
Population: 4-Fold rise in Menactra® vaccine antibodies were evaluated in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menactra® Booster Group | Group 2: Menactra® Primary Vaccine (Control) Group
Number analyzed (Participants) | 140 | 81
Percentage of Participants
  Serogroup A | 94 | 94
  Serogroup C | 84 | 90
  Serogroup Y | 97 | 98
  Serogroup W-135 | 99 | 100

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for up to 28 days post-vaccination
Arm/Group | Group 1: Menactra® Booster Group | Group 2: Menactra® Primary Vaccine (Control) Group
Serious Adverse Events (participants affected / at risk) | 1/151 | 0/85
Other Adverse Events (participants affected / at risk) | 32/151 | 15/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Menactra® Booster Group (N=151) | Group 2: Menactra® Primary Vaccine (Control) Group (N=85)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infections (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Menactra® Booster Group (N=151) | Group 2: Menactra® Primary Vaccine (Control) Group (N=85)
Injection site pain (General disorders) | 32 (32) | 15 (15)
Injection site erythema (General disorders) | 10 (10) | 8 (8)
Injection site swelling (General disorders) | 11 (11) | 8 (8)
Pyrexia (General disorders) | 16 (16) | 8 (8)
Headache (Nervous system disorders) | 13 (13) | 5 (5)
Malaise (General disorders) | 18 (18) | 11 (11)
Myalgia (General disorders) | 21 (21) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications